CLINICAL TRIAL: NCT04201977
Title: Comparison of Different Forms of Recovery on the Functionality After Physical Exercise: Randomized Clinical Trial
Brief Title: Comparison of Different Forms of Recovery on the Functionality After Physical Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Santa Maria (Other)
Responsible Party: Principal Investigator, Luis Ulisses Signori, Coordinator of the Postgraduate Program in Functional Rehabilitation, Universidade Federal de Santa Maria
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: nº 047670
Record Dates: First submitted 2019-12-10; First posted 2019-12-17 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-04

CONDITIONS: Massage; Inflammatory Response; Muscle, Skeletal; Cryotherapy Effect; Functional Disturbance
MeSH Terms: interventions — Exercise; Immersion; Cryotherapy

STUDY DESIGN:
Intervention Model Description: The four interventions will be randomized.
Who Masked: Outcomes Assessor
Masking Description: Evaluators will be blind to interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Exercise session followed passive recovery (Active Comparator): Prior each to the exercises sessions (4), volunteers will undergo specific warm-up in each exercise adopted (a series of 15 repetitions with 40% of the maximum load obtained in the 10RM test). The exercise sessions will consist of four sets for 10RM, with an interval of one minute between sets and two minutes between exercises. The exercise sequence (extension chair, squat and leg press) will be randomized through a closed brown envelope draw. Prior to the 10RM test and data collection, standardized instructions regarding the experimental procedure and exercise technique will be provided. Verbal stimuli to the volunteer will be performed during the evaluations and exercises (TEIXEIRA et al., 2014a, 2014b). The interval between each exercise session will be one week. Volunteers will not perform any form of recovery for 20 min after resistance exercise session (TEIXEIRA et al., 2014a, 2014b).
  Interventions: Other: Passive recovery
- Exercise session followed active recovery (Active Comparator): The interval between each exercise session will be one week. Prior each to the exercises sessions (4), volunteers will undergo specific warm-up in each exercise adopted (a series of 15 repetitions with 40% of the maximum load obtained in the 10RM test). The exercise sessions will consist of four sets for 10RM, with an interval of one minute between sets and two minutes between exercises. The exercise sequence (extension chair, squat and leg press) will be randomized through a closed brown envelope draw. Prior to the 10RM test and data collection, standardized instructions regarding the experimental procedure and exercise technique will be provided. Verbal stimuli to the volunteer will be performed during the evaluations and exercises (TEIXEIRA et al., 2014a, 2014b). Active recovery for 20 minutes (MIKA et al., 2016; CRISAFULLI et al., 2003; FAIRCHILD et al., 2003; VANDERTHOMMED; MAKROF; DEMOULIN, 2010);
  Interventions: Other: Active recovery
- Exercise session followed immersion in cold water recovery (Active Comparator): The interval between each exercise session will be one week. Prior each to the exercises sessions (4), volunteers will undergo specific warm-up in each exercise adopted (a series of 15 repetitions with 40% of the maximum load obtained in the 10RM test). The exercise sessions will consist of four sets for 10RM, with an interval of one minute between sets and two minutes between exercises. The exercise sequence (extension chair, squat and leg press) will be randomized through a closed brown envelope draw. Prior to the 10RM test and data collection, standardized instructions regarding the experimental procedure and exercise technique will be provided. Verbal stimuli to the volunteer will be performed during the evaluations and exercises (TEIXEIRA et al., 2014a, 2014b). Volunteers will be immersed in cold water immediately after exercise protocol (MACHADO et al., 2016b; MCDERMOTT et al., 2009).
  Interventions: Other: Immersion in cold water
- Exercise session followed foam roller recovery (Active Comparator): The interval between each exercise session will be one week. Prior each to the exercises sessions (4), volunteers will undergo specific warm-up in each exercise adopted (a series of 15 repetitions with 40% of the maximum load obtained in the 10RM test). The exercise sessions will consist of four sets for 10RM, with an interval of one minute between sets and two minutes between exercises. The exercise sequence (extension chair, squat and leg press) will be randomized through a closed brown envelope draw. Prior to the 10RM test and data collection, standardized instructions regarding the experimental procedure and exercise technique will be provided. Verbal stimuli to the volunteer will be performed during the evaluations and exercises (TEIXEIRA et al., 2014a, 2014b). Volunteers will undergo an FR session immediately after resistance exercise session (PEARCEY et al., 2015).
  Interventions: Other: Foam Roller Recovery

INTERVENTIONS:
Other: Foam Roller Recovery — Myofascial self-release will be developed through the foam roller (FR), where participants will use a custom-made foam roller constructed from a hollow polyvinyl chloride tube that will have an outside diameter of 10cm and a thickness of 0.5cm and will be surrounded by neoprene foam with a thickness of 1cm. Each volunteer will be shown the technique for the 5 muscle groups involved and the technique used for each muscle group. FR will consist of 45s of rolling for each muscle in the left lower extremity, 15s of rest, 45s in the lower right extremity. They will be instructed to begin with the practice on the most distal portion of the muscle. They will be instructed to place as much tolerable body mass on the FR at all times and to roll their body mass back and forth along the roller as smoothly as possible at a rate of 50 beats per minute (ie , 1 rolling motion for 1 to 2s). The total technique time is estimated at 10 to 15min (PEARCEY et al., 2015).
  Other Names: Self-massage; Foam Roller
  Arms: Exercise session followed foam roller recovery
Other: Active recovery — Active recovery for 20 minutes (MIKA et al., 2016) will consist of pedaling on a stationary bike at a speed of 50 to 60 rpm. The load (49 ± 9 W) will be adjusted individually so that the heart rate is close to 100 bpm (about 50% of the theoretical maximum heart rate). This effort intensity is similar to that used in the literature (CRISAFULLI et al., 2003; FAIRCHILD et al., 2003; VANDERTHOMMED; MAKROF; DEMOULIN, 2010)
  Other Names: Exercise
  Arms: Exercise session followed active recovery
Other: Immersion in cold water — Immersion in cold water will consist of the individual sitting in a plastic pool with water at the water level of the umbilical scar. Water temperature is between 11 and 15ºC, for a period between 10 and 15 minutes immediately after the exercise protocol (MACHADO et al., 2016b; MCDERMOTT et al., 2009). Water temperature will be controlled by adding or removing ice. This method has been applied by studies conducted by our research group (MISSAU; SIGNORI, 2017).
  Other Names: Cryotherapy
  Arms: Exercise session followed immersion in cold water recovery
Other: Passive recovery — Volunteers will be seated for 20 min after the resistance exercise session (TEIXEIRA et al., 2014a, 2014b).
  Other Names: Control
  Arms: Exercise session followed passive recovery

SUMMARY:
Delayed onset muscle soreness (DOMS) and decrease of musculoskeletal function are due to high intensity training and / or sports activities. These occur due to micro lesions of muscle tissue resulting in nociceptor sensitization. Non-pharmacological interventions to attenuate DOMS and favor muscle recovery have been studied. These interventions aim to maintain performance levels, especially in competitions. Among these interventions, cryotherapy (cold water immersion) and active recovery already have good clinical evidence. Currently a new proposal has been gaining ground for myofascial self-release (foam roller), however its mechanisms and clinical evidence are not yet well established. The aim of the present research is to compare the effects of passive recovery, active recovery, cold water immersion recovery and recovery through myofascial self-release on DOMS and the functionality of healthy volunteers undergoing resistance exercise.

DETAILED DESCRIPTION:
The volunteers included in the study will perform an evaluation to verify the eligibility criteria, physical evaluation (weight, height, systemic blood pressure) and functional capacity to determine the exercise parameters. After will be presented to the four interventions, ie the recovery techniques after the exercises favoring their adaptation. There will be four resistance exercise sessions followed by interventions with a one week interval between each session. Interventions (passive recovery = 1, active recovery = 2, recovery with IAF = 3 and recovery with myofascial self-release = 4) will be randomized. Functionality assessments will be performed before and one hour after the intervention protocol. DOMS will be evaluated 24 and 72 hours after the exercise protocol. Evaluators will be blind to interventions.

ELIGIBILITY:
Inclusion Criteria:

* Male,
* Literate,
* Normotensive volunteers,
* Aged minimum18 to maximum 35 years old,
* Physically active (IPAQ scale).
* Body mass index (BMI: kg / m2) greater than 30

Exclusion Criteria:

* Use of food supplements and medication
* Consume alcoholic beverages (+ once a week)
* Present of musculoskeletal disorders,
* Previous diagnosis of diseases (rheumatologic, cardiovascular diseases, as well as neurological, oncological, immunological and hematological diseases)
* Psychiatric and / or cognitive problems.

On the day of the exams will be excluded:

* Volunteers who present symptoms of musculoskeletal disorders,
* Consume ergogenic substances (24h),
* Consume alcoholic beverages and foods containing alcohol or caffeine (24h)
* Have performedintense physical activities 72 hours before the exam.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Isometric peak torque | 30 minutes after the interventions
  Isometric peak torque will be measured by a load cell of a tensile-compression dynamometer (EMGSystem, São José dos Campos, Brazil), with a capacity of 500 Kgf and a resolution of 0.1 kg, a set of fixing cables, a A/D converter board (EMGSystem, São José dos Campos, Brazil), connected to a computer and analyzed by the software EMGSystem Lab V1.2_ 2010. For each muscle group, a minimum of 4 and a maximum of 10 measurements of each movement will be performed. This variation in the number of measurements is so that the last measurement is not the highest value during the test and so that the three highest values differ by less than 5%. For analysis will be considered the highest value (NELLESSEN et al., 2015). During the evaluations, standardized and vigorous verbal encouragement will be performed during the maneuver, with the aim of stimulating the individual to exert maximum effort during the entire muscle contraction time.Data will be presented in kgf.

SECONDARY OUTCOMES:
Subjective exertion perception | 30 minutes after the interventions
  Subjective exertion perception ny the Borg scale (FOSTER et al. 2001). The scale ranges from 0 (no pain) to 10 (maximum bearable pain). Data will be presented in points average.
Flexibility | 30 minutes after the interventions
  The flexibility will be assessed by the Bank of Wells and Dilon (SIGNORI et al., 2008) and Lunge Test (CHISHOLM et al. 2012). Data will be presented in centimeter (cm).
Muscle power | 30 minutes after the interventions
  Muscle power will be assessed by single-limb general function (Single Hop Test) (BOLGLA; KESKULA, 1997). Data will be presented in centimeter (cm).
Agility | 30 minutes after the interventions
  Agility will be assessed by t-test (LATORRE ROMÁN ; VILLAR MACIAS; GARCÍA PINILLOS, 2017). Data will be presented in seconds (s)
Speed | 30 minutes after the interventions
  Speed will be evaluated by 30-meter test (PEARCEY et al., 2015). Data will be presented in seconds (s).
Muscle endurance | 30 minutes after the interventions
  Muscle fatigue strength will be assessed by the sit-up test (TVETER et al., 2014). Data will be presented by the number of repetitions.
Systemic blood pressure | 60 minutes after the interventions
  Blood pressure (BP) monitoring (Systolic blood pressure - SBP, Diastolic Blood Pressure - DBP and Mean Blood Pressure - MBP) will be performed using a multiparametric monitor (Dixtal, model 2021, Manaus, Brazil). The cuff will be positioned on the right arm with the patient positioned in the supine position on the stretcher. Data will be presented in mmHg.
Heart rate variability | 60 minutes after the interventions
  Heart rate variability (HRV) will be assessed before exercise and after interventions. The autonomic balance will be evaluated by the HRV, for the acquisition of the signal will be used a Polar frequency pulse model 810i (GAMELIN; BERTHOTOIN; BOSQUET, 2016). The acquisition of the electromyographic signal (ECG sampling rate - 1 kHz) of the RR interval time series will be acquired by continuous interval and will occur before and immediately after the interventions. For data collection the volunteer will remain lying supine at rest for 10 minutes and after standing for the same period of time, after the procedure will be repeated with breath control (16 movements per minute; I / E: 2 / 3) (NARDI et al., 2017). The analysis will be done by spectral power density (European Society of Cardiology & The North American Society of Pacing and Electrophysiology, 1996). Data will be presented absolute units (ms2) and your normalized units (n.u.).
Delayed onset muscle soreness | DOMS will be evaluated 24, 48 and 72 hours after the exercise protocol.
  Delayed onset muscle soreness (DOMS) will be evaluated by visual analog scale (EVA). The scale ranges from 0 (no pain) to 10 (maximum bearable pain).

CONTACTS AND LOCATIONS:
Locations (1):
- Luis Ulisses Signori, Santa Maria, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No
After publication of the results, the data will be made available to any researcher who requests via email.

REFERENCES:
- [Background] Machado AF, Almeida AC, Micheletti JK, Vanderlei FM, Tribst MF, Netto Junior J, Pastre CM. Dosages of cold-water immersion post exercise on functional and clinical responses: a randomized controlled trial. Scand J Med Sci Sports. 2017 Nov;27(11):1356-1363. doi: 10.1111/sms.12734. Epub 2016 Jul 19. PMID 27430594
- [Background] Latorre Roman PA, Villar Macias FJ, Garcia Pinillos F. Effects of a contrast training programme on jumping, sprinting and agility performance of prepubertal basketball players. J Sports Sci. 2018 Apr;36(7):802-808. doi: 10.1080/02640414.2017.1340662. Epub 2017 Jun 21. PMID 28636435
- [Background] Tveter AT, Dagfinrud H, Moseng T, Holm I. Health-related physical fitness measures: reference values and reference equations for use in clinical practice. Arch Phys Med Rehabil. 2014 Jul;95(7):1366-73. doi: 10.1016/j.apmr.2014.02.016. Epub 2014 Mar 5. PMID 24607837
- [Result] Mika A, Oleksy L, Kielnar R, Wodka-Natkaniec E, Twardowska M, Kaminski K, Malek Z. Comparison of Two Different Modes of Active Recovery on Muscles Performance after Fatiguing Exercise in Mountain Canoeist and Football Players. PLoS One. 2016 Oct 5;11(10):e0164216. doi: 10.1371/journal.pone.0164216. eCollection 2016. PMID 27706260
- [Result] Crisafulli A, Orru V, Melis F, Tocco F, Concu A. Hemodynamics during active and passive recovery from a single bout of supramaximal exercise. Eur J Appl Physiol. 2003 Apr;89(2):209-16. doi: 10.1007/s00421-003-0796-4. Epub 2003 Mar 4. PMID 12665987
- [Result] Fairchild TJ, Armstrong AA, Rao A, Liu H, Lawrence S, Fournier PA. Glycogen synthesis in muscle fibers during active recovery from intense exercise. Med Sci Sports Exerc. 2003 Apr;35(4):595-602. doi: 10.1249/01.MSS.0000058436.46584.8E. PMID 12673142
- [Result] Vanderthommen M, Makrof S, Demoulin C. Comparison of active and electrostimulated recovery strategies after fatiguing exercise. J Sports Sci Med. 2010 Jun 1;9(2):164-9. eCollection 2010. PMID 24149681
- [Result] McDermott BP, Casa DJ, Ganio MS, Lopez RM, Yeargin SW, Armstrong LE, Maresh CM. Acute whole-body cooling for exercise-induced hyperthermia: a systematic review. J Athl Train. 2009 Jan-Feb;44(1):84-93. doi: 10.4085/1062-6050-44.1.84. PMID 19180223
- [Result] MISSAU, E.; SIGNORI, L. U. Imersão na água fria na resposta inflamatória após exercícios resistidos. Revista Brasileria de Medina do Esporte, v. In submiss, 2017.
- [Result] Pearcey GE, Bradbury-Squires DJ, Kawamoto JE, Drinkwater EJ, Behm DG, Button DC. Foam rolling for delayed-onset muscle soreness and recovery of dynamic performance measures. J Athl Train. 2015 Jan;50(1):5-13. doi: 10.4085/1062-6050-50.1.01. Epub 2014 Nov 21. PMID 25415413
- [Result] TEIXEIRA, A. D. O. et al. Inflammatory response after session of resistance exercises in untrained volunteers. Acta Scientiarum. Health Sciences, v. 37, n. 1, p. 31-39, 2014a.
- [Result] TEIXEIRA, A. D. O. et al. The importance of adjustments for changes in plasma volume in the interpretation of hematological and inflmmatory responses after resistance exercise. Journal of Exercise Physiology, v. 17, n. 4, p. 72-83, 2014b.
- [Result] Nellessen AG, Donaria L, Hernandes NA, Pitta F. Analysis of three different equations for predicting quadriceps femoris muscle strength in patients with COPD. J Bras Pneumol. 2015 Jul-Aug;41(4):305-12. doi: 10.1590/S1806-37132015000004515. PMID 26398750
- [Result] Foster C, Florhaug JA, Franklin J, Gottschall L, Hrovatin LA, Parker S, Doleshal P, Dodge C. A new approach to monitoring exercise training. J Strength Cond Res. 2001 Feb;15(1):109-15. PMID 11708692
- [Result] Chisholm MD, Birmingham TB, Brown J, Macdermid J, Chesworth BM. Reliability and validity of a weight-bearing measure of ankle dorsiflexion range of motion. Physiother Can. 2012 Fall;64(4):347-55. doi: 10.3138/ptc.2011-41. PMID 23997389
- [Result] Bolgla LA, Keskula DR. Reliability of lower extremity functional performance tests. J Orthop Sports Phys Ther. 1997 Sep;26(3):138-42. doi: 10.2519/jospt.1997.26.3.138. PMID 9276854
- [Result] SIGNORI, L. U. et al. Efeito de agentes térmicos aplicados previamente a um programa de alongamentos na flexibilidade dos músculos isquiotibiais encurtados. Revista Brasileira de Medicina do Esporte, v. 14, n. 4, p. 328-331, 2008.
- [Result] Giles D, Draper N, Neil W. Validity of the Polar V800 heart rate monitor to measure RR intervals at rest. Eur J Appl Physiol. 2016 Mar;116(3):563-71. doi: 10.1007/s00421-015-3303-9. Epub 2015 Dec 26. PMID 26708360
- [Result] NARDI, A. T. DE et al. Different frequencies of transcutaneous electrical nerve stimulation on sympatho-vagal balance. Acta Scientiarum. Health Sciences, v. 39, n. 1, p. 9, 2017.
- [Result] Heart rate variability. Standards of measurement, physiological interpretation, and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. Eur Heart J. 1996 Mar;17(3):354-81. No abstract available. PMID 8737210
- [Derived] Arbiza BCC, da Silva AMV, de Lima KS, Rubin Neto LJ, Nunes GS, Jaenisch RB, Puntel GO, Signori LU. Effect of foam rolling recovery on pain and physical capacity after resistance exercises: A randomized crossover trial. J Bodyw Mov Ther. 2024 Jan;37:226-232. doi: 10.1016/j.jbmt.2023.11.022. Epub 2023 Nov 19. PMID 38432810